CLINICAL TRIAL: NCT06685003
Title: Phase II: Scalable Digital Delivery of Evidence-based Training for Addiction Professionals to Maximize Treatment Admission and Retention Rates of Opioid Use Disorder in Affected Families
Brief Title: Phase II: Scalable Digital Delivery of CRAFT Training for Professionals to Maximize Treatment Rates of OUD in Families
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: We The Village, Inc. (Other)
Collaborators: Public Health Management Corporation (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2403; 4R44DA053845-02 (NIH)
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Community Reinforcement And Family Training; Family Health; Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Conduct a fully randomized controlled trial of 3 levels of digital training (Level 1 - Digital tutorial only [T]; Level 2 - Tutorial & digital training materials for self-study [TM]; Level 3 - Tutorial, digital materials, feedback and coaching [TMC]) to examine the effects of training on CRAFT knowledge, fidelity, and treatment entry and retention.
Who Masked: Outcomes Assessor
Masking Description: The participants will know what group they are in. When data is sent to the statistician for analysis it will be coded in the groups (e.g., 123) without informing which is which. This masks (or blinds) him to the condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- T - Digital Tutorial overview (Active Comparator): A digital tutorial consisting of a curriculum dashboard for review of 20 modules, including videos, PDFs, text and quizzes, which are to be unlocked sequentially over seven weeks. Modules remain available during the 6-month study timeframe. Participants receive weekly contact encouraging engagement in all of the materials available to them.
  Interventions: Behavioral: Digital Tutorial overview
- TM - Digital Tutorial plus training Materials (Experimental): Participants receive the digital tutorial (T), plus access to 15 additional in depth modules of digital training materials also released weekly alongside the tutorial modules. Modules remain available during the 6-month study timeframe. Participants receive weekly contact encouraging engagement in all of the materials available to them.
  Interventions: Behavioral: Digital Tutorial overview; Behavioral: Digital Tutorial plus training Materials
- TMC - Digital Tutorial plus training Materials plus feedback and Coaching (Experimental): Participants receive the digital tutorial (T) plus the digital Training materials (TM), plus they submit audio recordings of sessions with clients and receive feedback on their application of CRAFT and receive group coaching on how to improve.
  Interventions: Behavioral: Digital Tutorial overview; Behavioral: Digital Tutorial plus training Materials; Behavioral: Digital Tutorial plus training Materials plus feedback and Coaching

INTERVENTIONS:
Behavioral: Digital Tutorial overview — Self study of a digital tutorial covering an overview of CRAFT designed to be reviewed within 7 weeks and revisited over 6 months.
  Other Names: T
Behavioral: Digital Tutorial plus training Materials — Self study of a digital tutorial covering an overview of CRAFT and deeper materials designed to be reviewed within 7 weeks and revisited over 6 months.
  Other Names: TM
  Arms: TM - Digital Tutorial plus training Materials; TMC - Digital Tutorial plus training Materials plus feedback and Coaching
Behavioral: Digital Tutorial plus training Materials plus feedback and Coaching — Self study of a digital tutorial covering an overview of CRAFT and deeper materials designed to be reviewed within 7 weeks and revisited over 6 months. Plus group coaching and feedback on audio recordings of CRAFT procedures used in sessions
  Other Names: TMC
  Arms: TMC - Digital Tutorial plus training Materials plus feedback and Coaching

SUMMARY:
The goal of this project is to demonstrate digital training efficacy at scale and commercial readiness.

This pilot project will advance piloted digital training programs for CRAFT and maximize scalability. In this project, investigators will:

Aim 1: Optimize the digital CRAFT training product based on data and feedback from the pilot and commercialization advisors.

Aim 2: Conduct a fully powered randomized control trial of 3 levels of digital training (Level 1 - Digital tutorial only [T]; Level 2 - Tutorial & digital training materials for self-study [TM]; Level 3 - Tutorial, digital materials, feedback and coaching [TMC]) to examine the effects of training on CRAFT knowledge, fidelity, and plus IP treatment entry/retention and counselor skill pre- and post-tutorial, at 12 weeks and at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Be over 19
* Live in the US
* Work in a counselor-related profession
* Have counseling work that involves clients
* Work with CSOs impacted by OUD, or could work with this type of client
* Have not been certified in CRAFT
* Have not participated in the 2023 WTV counselor training pilot study
* Be able to provide at least 45-minute individual counselor sessions to at least one CSO (CSO)
* Be able and willing to complete intervention activities over the course of the 12-week study as determined by the random assignment including: participating in the tutorial and training and submitting the required session audiotapes
* Report having access to a computer and smartphone with internet access, email, and word processing capability
* Demonstrate complete understanding of the requirements for participation in the study by reading and signing the consent form and completing the online consent quiz or confirmation call
* Provide valid locator information to allow research and CRAFT training staff to contact them to schedule study-related appointments
* Complete the first assessment mock session with our standardized patient (SP) and pre-tutorial surveys

Exclusion Criteria:

* Does not agree to participate
* Does not complete the baseline assessment requirements
* Is not English-speaking
* Participated in the Qualitative Review aspect of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-11-04 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
CRAFT Procedure Fidelity | 3 months, 6 months
  CRAFT performance on the mock sessions observed by trained coders rating performance of each CRAFT treatment entry procedure (6 items), homework procedures (2 items), overall CRAFT approach (2 items), and general clinical skill (4 items) on a 5-point scale (i.e., 1 =poor; 3 =satisfactory; 5 =excellent). Total score will be calculated across all 14 items for each participant. Average scores on each procedure and in total will be calculated for each participant group at baseline and at follow-ups. Scores can range from 6 - 30 on treatment entry; 2 - 10 on homework and CRAFT approach; 4 - 20 on general clinical skill; and 14 - 70 on the overall total.

SECONDARY OUTCOMES:
3 months | 3 months, 6 months
  Measuring the proficiency with which participants answer questions about the CRAFT approach.
  Measuring the proficiency with which participants answer questions about the CRAFT approach.
  The 20-item CRAFT Knowledge Test is scored by calculating the number of correct answers for each individual and then averaging scores across participants within each group (T, TM, TMC). Scores could range from 0 - 20.
Program Implementation Potential Scale | 3 months, 6 months
  Measured by program implementation potential questionnaire containing 25 Items; responses on 1-6 scale (strongly agree to strongly disagree).

OTHER OUTCOMES:
New Treatment Entry: Identified Patient Treatment Entry Status | 3 months, 6 months
  Participants report whether their client's loved one has attended any treatment for their opioid use problem since the baseline assessment by answering questions regarding participation in treatment. In addition, reports of treatment entry to WTV staff were categorized as treatment entry. The outcome is the proportion of participants reporting that their client's loved one (identified patient; IP) entered new treatment

CONTACTS AND LOCATIONS:
Locations (1):
- We The Village, Inc., New York, New York, United States

IPD SHARING:
Plan to Share IPD: No